CLINICAL TRIAL: NCT04484350
Title: Blood Pressure Management in Stroke Following Endovascular Treatment
Acronym: DETECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DETECT-v1.0
Record Dates: First submitted 2020-07-06; First posted 2020-07-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute; Vessels; Occlusion; Blood Pressure; Endovascular Thrombectomy; Mechanical Thrombectomy
Keywords: endovascular stroke treatment; successful recanalization; transcranial Doppler Ultrasound; intracranial hemorrhage
MeSH Terms: conditions — Stroke; Bites and Stings; Intracranial Hemorrhages | interventions — Labetalol; Hydralazine; Enalapril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Blood Pressure management (Experimental): Participants assigned to the intensive blood pressure management arm will be treated using approved antihypertensive medications to have systolic blood pressure readings under 140 mmHg for the first 48 hours after enrollment into the study.
  Interventions: Drug: Labetalol; Drug: Hydralazine; Drug: Enalapril
- Standard Blood Pressure management (Active Comparator): Participants assigned to the standard blood pressure management arm will be treated using approved antihypertensive medications to have systolic blood pressure readings under 180 mmHg for the first 48 hours after enrollment into the study.
  Interventions: Drug: Labetalol; Drug: Hydralazine; Drug: Enalapril

INTERVENTIONS:
Drug: Labetalol — 10 - 20 mg IV q15 minutes PRN until systolic BP below target (max 300 mg per 24 hours)
Drug: Hydralazine — 10 - 20 mg IV bolus q20 min until systolic BP below target (max 240 mg per 24 hours)
Drug: Enalapril — 1.25 - 2.5 mg IV bolus and then q6h PRN.

SUMMARY:
The aim of DETECT is to prove the feasibility of a multicenter phase III trial testing the hypothesis that intensive blood pressure control immediately after successful endovascular stroke thrombectomy can improve patient outcomes. Patients with stroke who have ongoing high blood pressure after successful clot retrieval will be included. Participants will be randomly placed (like flipping a coin) in one of two groups. There will be a 50% chance of each patient being placed to either group. The first group will be allowed to have a higher blood pressure range that is consistent with current recommendations. The second group will be given medications to bring their blood pressure down into a normal range. These blood pressure targets will be maintained for 48 hours. We will collect patient brain images and levels of stroke disability up to 90 days after their clot retrieval.

DETAILED DESCRIPTION:
Current guidelines from the American Heart Association/ American Stroke Association (AHA/ ASA) propose thresholds of systolic blood pressure (BP) less than 180 mm Hg and diastolic BP less than 105 mm Hg during and for the first 24 hours following endovascular treatment (EVT), which have been arbitrarily inherited from previous intravenous thrombolysis guidelines. Although there is plethora of evidence from observational cohort studies suggesting that increased BP following EVT is associated with higher likelihood of both intracranial hemorrhage and unfavorable clinical outcomes, the potential for residual confounding in these observational datasets limits their interpretation. The blooD prEssure management in sTroke following EndovasCular Treatment (DETECT) trial is a single-center, pragmatic, pilot, prospective open label, blinded end point, randomized controlled trial testing the hypothesis that intensive BP management following successful EVT is feasible. The primary objective of DETECT is to determine the feasibility of a RCT assessing the efficacy and safety of intensive BP lowering compared to standard of care in rates of hemorrhagic transformation and functional outcome following successful EVT in acute ischemic stroke patients with large vessel occlusion. We will include adult patients with acute ischemic stroke achieving successful reperfusion (TICI more or equal to 2b) of a proximal large vessel occlusion in the anterior circulation after EVT. Eligible patients will be randomized 1:1 within 60 minutes from the end of the EVT procedure to either intensive (systolic BP target <140 mmHg) or standard BP management (systolic BP target <180 mmHg) for the first 48 hours after randomization. Patients with presence of concomitant ipsilateral or contralateral extracranial vessel occlusion or remaining stenosis ≥80% after the end of the EVT, and/or patients having any medical condition where randomization to either standard or intensive BP lowering would not be acceptable at the discretion of the treating physician will be excluded from participating. The trial will be embedded within an established national EVT registry that focuses on improving quality of management of patients receiving EVT for ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18 years.
* Eligible for endovascular treatment (EVT) within 24 hours from symptom onset according to current clinical practice.
* Presence of a proximal large vessel occlusion in the anterior circulation, defined as occlusion of the intracranial segment of the internal carotid artery and/or occlusion of the M1 segment or proximal M2 segment of the middle cerebral artery.
* Successful recanalization after the end of the EVT procedure, defined as modified thrombolysis in cerebral ischemia (mTICI) score equal or more than 2b.
* Sustained elevated systolic BP level after recanalization, defined as 2 consecutive systolic BP readings ≥ 150 mmHg (or ≥ 140 mmHg if the participant has a known history of hypertension) taken more than 5 minutes apart.
* Ability of the patient or legal representative to provide informed consent.
* Randomization within 60 minutes from the end of the EVT procedure.

Exclusion Criteria:

* Presence of concomitant ipsilateral or contralateral extracranial vessel occlusion or remaining stenosis ≥80% after the end of the EVT.
* Symptomatic intracranial hemorrhage after the end of EVT procedure.
* Any medical condition where randomization to either standard or intensive BP lowering would not be acceptable at the discretion of the investigators and/or the treating physician.
* Pregnancy.
* Enrollment in another acute stroke therapeutic trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Mean enrollment rate. | through study completion, an average of 18 months
  The predefined target is to achieve a mean enrollment rate of 2 patients per month.
Number of participants with treatment allocation change. | 48 hours from treatment initiation
  The predefined target is that at least 80% of the participants remain within their assigned treatment group, and not changing treatment allocation for any reason.

SECONDARY OUTCOMES:
Number of participants with any intracranial hemorrhage. | 24±12 hours from treatment initiation
  As identified in the follow-up computed tomography scan.
Absolute difference in flow velocity measurements in transcranial Doppler. | 0-18 hours from treatment initiation
  Assessed with the adjusted mean flow velocities of the recanalized vessel on transcranial Doppler examination.
Absolute difference in the NIH Stroke Scale change at day 1. | 24±12 hours from treatment initiation
  NIH Stroke Scale ranges from 0 to 42, with higher scores indicating more severe impairment caused by a stroke.
Absolute difference in the NIH Stroke Scale change at day 2. | 48±12 hours from treatment initiation
  NIH Stroke Scale ranges from 0 to 42, with higher scores indicating more severe impairment caused by a stroke.

OTHER OUTCOMES:
Absolute difference in mean systolic blood pressure values. | 48 hours from treatment initiation
  Difference in mean systolic blood pressure values between the two arms.
Number of participants with symptomatic intracranial hemorrhage. | 24±12 hours from treatment initiation
  According to the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST), National Institute of Neurological Disorders and Stroke (NINDS) and European-Australian Cooperative Acute Stroke Study 2 (ECASS 2) definitions.
Number of deaths during hospitalization. | Day 7 from treatment initiation or hospital discharge
  All-cause in-hospital mortality.
Number of deaths during follow-up. | Day 90±10 from treatment initiation
  All-cause mortality.
Number of participants with neurological deterioration. | 24 hours from treatment initiation
  Defined as ≥4 points decline in the National Institute of Health Stroke Scale (NIHSS) from randomization or death.
Functional outcome during hospitalization. | Day 7 from treatment initiation or hospital discharge
  Ordinal shift analysis of the full range of category scores (0-6) of the modified Rankin Scale (mRS).
Functional outcome during follow-up. | Day 90±10 from treatment initiation
  Ordinal shift analysis of the full range of category scores (0-6) of the modified Rankin Scale (mRS).
Number of participants with favorable functional outcomes during hospitalization. | Day 7 from treatment initiation or hospital discharge
  Favorable functional outcomes defined as modified Rankin Scale (mRS) scores of 0-1 or 0-2.
Number of participants with favorable functional outcomes during follow-up | Day 90±10 from treatment initiation
  Favorable functional outcomes defined as modified Rankin Scale (mRS) scores of 0-1 or 0-2.
Absolute difference in the decline of the Alberta stroke program early CT scores. | 24±12 hours from treatment initiation
  The Alberta Stroke Program Early CT Score (ASPECTS) is a 10-point (range 0-10) quantitative topographic imaging scale with higher scores indicating more favorable imaging profiles. Differences will be assessed between the baseline and repeat computed tomography scan.
Absolute difference in final infarct volumes. | Day 7 from treatment initiation
  As assessed in the magnetic resonance imaging (MRI) scan, when available.
Absolute difference in hospital stay. | Day 7 from treatment initiation or hospital discharge
  Duration of hospital length of stay in days.

CONTACTS AND LOCATIONS:
Overall Officials: Aristeidis H Katsanos, MD, Principal Investigator — Hamilton General Hospital, Hamilton Health Sciences
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes